CLINICAL TRIAL: NCT02758743
Title: The Efficacy of Acetium Lozenges in Intervention for Smoking Cessation: A Double-blind, Placebo-controlled Trial
Brief Title: The Efficacy of Acetium Lozenges in Intervention for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biohit Oyj (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AL-SMOQUIT-2
Record Dates: First submitted 2016-04-21; First posted 2016-05-02 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Smoking Cessation
Keywords: smoking; tobacco; smoking cessation
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetium Lozenge (Experimental): Acetium lozenge (L-cysteine 3mg) is used in context of each cigarette smoked.
  Interventions: Drug: Acetium Lozenge
- Placebo (Placebo Comparator): Identical in appearance with Acetium lozenge, placebo lozenges will be used in the same manner as in experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetium Lozenge — Slow-release L-Cysteine to block smoke.derived acetaldehyde in saliva thereby inhibiting the formation of harmans
  Arms: Acetium Lozenge
Drug: Placebo — Placebo with no active substance will not have the effect on intervention device.
  Arms: Placebo

SUMMARY:
The purpose of this study is to validate the novel hypothesis that regular use of Acetium Lozenge is promising novel method to assist in smoking cessation.

The aim of this confirmatory study is to affirm the promising results obtained in a previous smoking intervention trial with Acetium lozenge. If successful, the trial gives adequate power to confirm, that the Acetium lozenge represents a breakthrough in the development of smoking intervention methods.

DETAILED DESCRIPTION:
Background: Smoking dependence has been traditionally ascribed to nicotine, the major psychoactive component of tobacco (nicotine addiction). Dependence on smoking, however, is a much more complex issue than just nicotine addiction, and during the past several decades, a wide variety of approaches have been used in intervention for smoking cessation, with variable success.

Tobacco smoke contains several classes of carcinogens, including acetaldehyde in high concentrations. Acetaldehyde from the tobacco smoke is easily dissolved into the saliva during smoking, and thus, toxic aldehydes could mediate the carcinogenic effect of tobacco smoke through the saliva. In 2009, IARC proclaimed acetaldehyde as Group I carcinogen, equivalent to asbestos, formaldehyde and others.

Based on observations that in rodents, acetaldehyde induces reinforcing effects acting in concert with nicotine, Talhout et al (2007) hypothesized that harmans (condensation products of acetaldehyde and biogenic amines) may be responsible for these nicotine-reinforcing effects of acetaldehyde. Harmans are formed in cigarette smoke, and blood harman levels among smokers appear to be 2-10 times higher than in non-smokers. Harmans inhibit monoamine oxidase (MAO), and like other MAO-inhibitors, these might help maintaining the behavioral sensitization to nicotine. This led these authors to speculate that acetaldehyde may increase the addictive potential of tobacco products via formation of harmans in cigarette smoke.

It has been known for several decades that L-cysteine (a nonessential amino acid) is able to eliminate the toxicity of acetaldehyde by reacting covalently with acetaldehyde to form a stable 2-methylthiazolidine-4-carboxylic acid (MTCA). This simple principle was used in the recent innovation of Biohit HealthCare's Acetium™ capsule containing 100mg L-cysteine. Oral administration of Acetium was confirmed to effectively bind acetaldehyde originated from ethanol metabolism in the stomach, raising the idea that L-cysteine could also be used to eliminate acetaldehyde dissolved into the saliva during smoking. Indeed, Salaspuro et al. (2006) confirmed that orally administered L-cysteine (5mg)-containing sucking tablet (lozenge) totally inactivated acetaldehyde in the saliva during smoking.

Given the above, it is tempting to speculate that elimination of acetaldehyde in the saliva during cigarette smoking by L-cysteine sucking tablets, might effectively block (or reduce) the formation of harmans, reduce their high blood levels, and thus alleviate the acetaldehyde-enhanced nicotine addiction (by reducing MAO-inhibition) among smokers. The present study is designed to validate the novel hypothesis that regular use of Acetium lozenges in context with smoking is an effective intervention for cessation of cigarette smoking.

Objective: To test the efficacy of Acetium lozenges (used simultaneously with smoking) to trigger the quit from cigarette smoking as compared with similarly administered placebo preparation.

Study design: A double-blind, placebo-controlled clinical trial comparing Acetium lozenges and placebo as triggers of cigarette smoking cessation during one-year intervention.

Methods: A cohort of 1.800 current cigarette smokers will be enrolled by public invitation. Eligible subjects must be current cigarette smokers (no limitation as to pack years), who are well motivated to refrain from smoking, and who give a written consent to participate. The subjects will be randomly allocated to two groups (n=900 in each), receiving either Acetium lozenges or placebo, in a double-blind setting, where both the examiners and the test subjects are blinded to the test substance. All subjects must consent for not using any other measures of smoking cessation intervention. All subjects are requested to fill in a structured questionnaire recoding their detailed smoking history and assessing their nicotine dependence by FTND (Fagerström Test for Nicotine Dependence) and breath CO-monitoring. The subjects will be administered a smoking diary, to be filled on daily basis, recording the daily numbers of cigarettes, test lozenges and subjective sensations of smoking. These diaries are returned to study monitors on three-monthly FU visits, when also subjected to new FTND and CO-monitoring.

The primary study endpoints include PPA (point prevalence of abstinent rate) and PA (prolonged abstinence), used for calculating OR (95%CI) between the two study arms by logistic regression. Changes in FTND score and CO-levels represent intermediate surrogate endpoints of PP and PA. In addition, time to quit (TTQ) and duration of quit (QT=quit time) can be used as dependent variables in univariate (Kaplan-Meier) and multivariate (Cox) survival analyses. GEE and Poisson models are used to estimate the covariates (Acetium/Placebo) of i) persistence of abstinence, and ii) quit events (events/person time at risk), respectively, based on multiple records (panel data) in a longitudinal setting. Finally, the predictors of the multiple outcomes in this intervention trial can be estimated using the novel competing-risks regression model, where i) no effect, ii) permanent quit, iii) temporary quit with relapse, and iv) smoking reduction, represent the competing-risks events.

The power of the study can be calculated specifically for each of these statistical techniques, most simply by the two-sample proportion test for PP and PA. This study (n=900 in both arms) is adequately powered (Type II error 0.80, type I error 0.05) to detect a true difference (in PP or PA) of 5% between the two arms, within the range of 10% vs. 20% quit rate in the two arms. Within this (10-20%) range, the study power is sensitive to any decrease in this difference, but allows less difference (7.5%) if the quit rate falls between 5% and 15% in the arms.

Specific aims: The null hypothesis of the study implicates that Acetium lozenges are not superior to placebo in the intervention for smoking quit during the 1-year intervention. Rejection or not of the null hypothesis is based on comparison of the two arms by the different statistical approaches listed above.

Impact of the study: This double-blind, placebo-controlled intervention trial will test the new hypothesis whether or not Acetium lozenges are superior to placebo as triggers of smoking quit when regularly used in context of smoking for a prolonged period. If this concept proves to be correct, the results will have a major clinical impact while providing an entirely novel approach to support regular smokers to withdraw this unhealthy habit.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years male/female
* current cigarette smoker
* motivated to quit smoking

Exclusion Criteria:

* serious smoking-related diseases
* pregnant and lactating women
* use of quit smoking medicine
* simultaneous participation in an other clinical trial
* earlier participation in the same trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1998 (Actual)
Dates: Start 2016-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Prolonged abstinence (PA), based on smoking diary | 6 months
  Prolonged abstinence, a sustained or continuous abstinence - is typically defined as not smoking for a period of several months after a quit attempt. Sometimes, this is for the entire period since the quit date, and sometimes it begins after an initial "grace or charm" period
Point prevalence of abstinence (PPA), based on smoking diary | 6 months
  Point prevalence is typically defined as not smoking on the day of follow-up (or for a few days before a follow-up day).

CONTACTS AND LOCATIONS:
Overall Officials: Kari Syrjänen, MD, PhD, Principal Investigator — Biohit Oyj
Locations (1):
- Kuulas Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
individual participants data not public.